CLINICAL TRIAL: NCT05073549
Title: Optimizing Antibiotic Use in Neonatal Intensive Care Units: A Collaborative Antimicrobial Stewardship Program in China
Brief Title: Optimizing Antibiotic Use in Neonatal Intensive Care Units in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: China Medical Board (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021144
Record Dates: First submitted 2021-09-06; First posted 2021-10-11 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Neonates

STUDY DESIGN:
Intervention Model Description: Pre- and post-study
  * The period from October 1st, 2019 to September 30th, 2021 will be used as the baseline period before the intervention. Clinical data of eligible infants in this period will be retrospectively collected from a previously established database of preterm infants.
  * The intervention will be initiated on October 1st, 2021. The period from October 1st, 2021 to September 31st, 2023 will be the intervention period and data will be prospectively collected.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collaborative antimicrobial stewardship group (Experimental): Collaborative antimicrobial stewardship intervention will be implemented in NICUs of this group.
  Interventions: Behavioral: Collaborative Antimicrobial Stewardship Program (ASP)

INTERVENTIONS:
Behavioral: Collaborative Antimicrobial Stewardship Program (ASP) — The collaborative ASP interventions will be implemented from October 1st, 2021 to September 30th, 2023 in all participating NICUs.
  The collaborative ASP interventions include two levels of interventions that will be delivered at the NICU level: the NICU-targeted ASP program and collaborative quality improvement interventions to facilitate implementation of the ASP.
  The core elements of the NICU-targeted ASP program include the establishment of ú ASP leader and team, development of the facility-specific antibiotic guidelines, checklist-led audit and feedback, and staff education.
  The collaborative quality improvement interventions include data feedback and benchmarking, a potential 'better practice' list on neonatal antibiotic use, implementation using Plan-Do-Study-Act cycles and collaborative learning.

SUMMARY:
This project aims to reduce antibiotic use in Chinese neonatal intensive care units (NICU) by 1) developing an adaptable framework of NICU-targeted antimicrobial stewardship programs (ASP); 2) implementing the NICU-targeted ASP in NICUs using a collaborative quality improvement method; and 3) evaluating the impact of ASP implementation on neonatal antibiotic use.

DETAILED DESCRIPTION:
Antibiotics overuse has been a critical problem in Chinese NICUs associated with the emerging antimicrobial resistance crisis. NICU-targeted ASP have rarely been implemented in Chinese NICUs. Collaborative quality improvement methods have been shown to facilitate clinical practice changes and improve outcomes.

In this two-year interventional pre-and post-study, a NICU-targeted ASP will be developed and implemented in Chinese NICUs using the collaborative quality improvement method. The investigators hypothesize that implementing the targeted ASP using a collaborative quality improvement method will reduce the overall antibiotic days of therapy by 20% over a two-year period, comparing the last year of intervention and the last year of baseline period before ASP implementation.

ELIGIBILITY:
Inclusion Criteria:

* All infants born at ≤31+6 weeks' gestation and admitted to the participating NICUs between October 1st, 2019 and September 30th, 2023.
* The period from October 1st, 2019 to September 30th, 2021 will be used as the baseline period before ASP intervention. Clinical data of eligible infants in this period will be retrospectively collected from a previously established database of preterm infants.
* The ASP implementation will be initiated on October 1st, 2021. The period from October 1st, 2021 to September 31st, 2023 will be the ASP intervention period and data will be prospectively collected.

Exclusion Criteria:

* Infants who are transferred to non-participating NICUs within 24 hours after birth.

Ages: 0 Days to 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10000 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Total antibiotic days of therapy (DOT) per 1000 patient-days | up to 180 days
  DOT is calculated as the sum of days of antibiotics used per patient.

SECONDARY OUTCOMES:
Total antibiotic days of therapy (DOT) per 1000 patient-days of third-generation cephalosporin | up to 180 days
  DOT is calculated as the sum of days of third-generation cephalosporin used per patient.
Total antibiotic days of therapy (DOT) per 1000 patient-days of fourth-generation cephalosporin | up to 180 days
  DOT is calculated as the sum of days of fourth-generation cephalosporin used per patient.
Total antibiotic days of therapy (DOT) per 1000 patient-days of piperacillin-tazobactam | up to 180 days
  DOT is calculated as the sum of days of piperacillin-tazobactam used per patient.
Total antibiotic days of therapy (DOT) per 1000 patient-days of carbapenem | up to 180 days
  DOT is calculated as the sum of days of carbapenem used per patient.
Total antibiotic days of therapy (DOT) per 1000 patient-days of vancomycin | up to 180 days
  DOT is calculated as the sum of days of vancomycin used per patient.
Total antibiotic days of therapy (DOT) per 1000 patient-days of linezolid | up to 180 days
  DOT is calculated as the sum of days of linezolid used per patient.
Incidence rate of infections caused by multi-resistant bacteria | up to 180 days
  Multi-resistant bacteria include carbapenem-resistant Enterobacter, methicillin-resistant Staphylococcus aureus, vancomycin-resistant Enterococcus, multi-resistant Acinetobacter, multi-resistant Pseudomonas aeruginosa.
Incidence rate of infections caused by multi-resistant bacteria | up to 180 days
  Multi-resistant bacteria include carbapenem-resistant Enterobacter, methicillin-resistant Staphylococcus aureus [MRSA], vancomycin-resistant Enterococcus [VRE], multi-resistant Acinetobacter, multi-resistant Pseudomonas aeruginosa.
Incidence rate of invasive fungal infections | up to 180 days
Incidence of mortality | up to 180 days
  Overall mortality and infection-related mortality
Incidences of major morbidities | up to 180 days
  Major morbidities include late-onset sepsis, necrotizing enterocolitis, bronchopulmonary dysplasia, retinopathy of prematurity and severe brain injury.
Length of hospital stay | up to 180 days

OTHER OUTCOMES:
Number of antibiotic courses initiated within 7 days after the discontinuity of the previous course | up to 180 days
  Safety measure which indicate insufficient antibiotic therapy.

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - Fujian Maternity and Child Health Hospital, Fuzhou, Fujian
  - Quanzhou Women and Children's Hospital, Quanzhou, Fujian
  - Gansu Provincial Maternity and Child Care Hospital, Lanzhou, Gansu
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Shenzhen Maternity and Child Health Care Hospital, Shenzhen, Guangdong
  - Women and Children's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Guizhou Women and Children's Hospital/Guiyang Children's Hospital, Guiyang, Guizhou
  - Henan Children's Hospital, Zhengzhou, Henan
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Children's Hospital, Changsha, Hunan
  - Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Suzhou Municipal Hospital affiliated to Nanjing Medical University, Suzhou, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Xining, Ningxia
  - Northwest Women's and Children's Hospital, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Qingdao Women and Children's Hospital, Qingdao, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Children' s Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Children's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Tianjin Obstetrics & Gynecology Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan